CLINICAL TRIAL: NCT03253666
Title: Nurses' Health Study and Health Professionals Follow-Up Study (Dermatological Component)
Status: Completed | Type: Observational
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Brown University (Other)
Responsible Party: Principal Investigator, Ashar Dhana, Research Associate, Harvard School of Public Health (HSPH)
Other Study IDs: CA186107
Record Dates: First submitted 2017-08-11; First posted 2017-08-18 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Skin Cancer; Melanoma; Non-melanoma Skin Cancer; Psoriasis; Rosacea; Lupus Erythematosus; Atopic Dermatitis
MeSH Terms: conditions — Skin Neoplasms; Melanoma; Psoriasis; Rosacea; Dermatitis, Atopic | interventions — Eating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nurses' Health Study: See "Detailed Description"
  Interventions: Other: Nutrient Intake
- Health Professionals Follow-Up Study: See "Detailed Description"
  Interventions: Other: Nutrient Intake

INTERVENTIONS:
Other: Nutrient Intake — Dietary nutrient intake (such as folate) and supplemental nutrient intake (such as folic acid)

SUMMARY:
To determine the relationships of dietary factors with the subsequent risk of dermatological diseases (such as skin cancers and inflammatory or autoimmune dermatoses) in a cohort of female registered nurses and male health professionals.

DETAILED DESCRIPTION:
The study population consisted of two ongoing cohorts: the Nurses' Health Study (NHS) and Health Professionals Follow-Up Study (HPFS). The NHS began in 1976 when 121,700 female nurses aged 33-55 years and residing in the United States responded to a baseline questionnaire. The HPFS began in 1986 when 51,529 male health professionals aged 40-75 years and residing in the United States completed a similar baseline questionnaire. Study investigators sent follow-up questionnaires biennially to participants to update information on past medical history as well as lifestyle factors.

Follow up was started in 1984 for the NHS and 1986 for the HPFS when diet was measured with an expanded food frequency questionnaire (FFQ). Participants in the NHS responded to an ~130 item semi-quantitative FFQ in 1984, 1986, and then every four years thereafter, while those in the HPFS responded to a similar FFQ in 1986 and then every four years thereafter. The FFQ collected information on average intake of each food item over the past year. It also specified a common serving size for each item. Participants could select from one of nine intake frequency choices, ranging from less than once per month to six or more times per day. Participants also provided information on current use and dose of multivitamins and use of other vitamin supplements.

For both cohorts, investigators repeatedly collected and updated information on several anthropometric and lifestyle factors such as weight, smoking status, alcohol use, coffee intake, and physical activity level. Information was also collected on several major risk factors for skin disease such as family history of melanoma, number of arm moles, natural hair color, sunburn susceptibility as a child or adolescent, number of lifetime blistering sunburns, type of tan after repeated sun exposure as a child or adolescent, and cumulative ultraviolet flux since baseline.

Study subjects reported new diagnoses biennially. After obtaining permission from participants, their medical and pathological records were acquired. Study physicians blinded to questionnaire information reviewed these records to confirm diagnoses

The study was approved by the institutional review boards of both Brigham and Women's Hospital and Harvard T.H Chan School of Public Health.

ELIGIBILITY:
Inclusion Criteria:

-Participants of these two cohorts

Exclusion Criteria:

* Participants with missing data on dietary intake at baseline
* Participants with a prior history of cancer (except non-melanoma skin cancer)
* For skin cancer, non-white participants because of low risk of skin cancer (such as melanoma) and small numbers.
* For melanoma, participants with in-situ melanomas, which comprise tumours restricted to the epidermis of the skin.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: See "Detailed Description"
Sampling Method: Probability Sample
Enrollment: 173229 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-05 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Multiple skin diseases | Skin disease/cancer [ NHS: Time Frame: 1984 - 2010 ] [ HPFS: Time Frame: 1986 - 2010 ]. Person time contribution from date of return of questionnaire to date of first report of skin disease/death/end of follow-up (whichever came first)
  Includes skin cancer, psoriasis, and other inflammatory and autoimmune skin diseases.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Li WQ, Cho E, Weinstock MA, Mashfiq H, Qureshi AA. Epidemiological Assessments of Skin Outcomes in the Nurses' Health Studies. Am J Public Health. 2016 Sep;106(9):1677-83. doi: 10.2105/AJPH.2016.303315. Epub 2016 Jul 26. PMID 27459457
- See also: Nurse's Health Study — http://www.nurseshealthstudy.org/